CLINICAL TRIAL: NCT00393627
Title: Efficacy of Behavioral Interventions to Improve Sleep in Adult Family Homes
Brief Title: Behavioral Sleep Intervention in Adult Family Homes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Sue McCurry, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24091-G; 03-7612-G 04
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Dementia
Keywords: Dementia; Sleep disturbance; Behavioral strategies; Alzheimer's Disease; Adult Family Homes
MeSH Terms: conditions — Dementia; Parasomnias; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sleep Education Program: The Sleep Education Program (SEP) is conducted by a licensed MS- or PhD-level mental health professional experienced in working with persons with dementia and their caregivers. The therapist meets with the AFH owner/operator and staff for four weekly sessions at the AFH. The SEP content includes information about the causes of sleep problems in dementia, and provides staff with assistance in developing customized resident behavioral sleep plans focused on environmental (light and noise), dietary (eliminating caffeine and excessive nighttime fluids), and sleep scheduling (reducing afternoon/ evening napping; consistent, appropriate bed and rising times) factors that are commonly associated with resident nighttime awakenings. A written manual is used.
  Interventions: Behavioral: Sleep Education Program
- 2 (Placebo Comparator): Routine medical care
  Interventions: Behavioral: Sleep Education Program

INTERVENTIONS:
Behavioral: Sleep Education Program — The Sleep Education Program (SEP) is conducted by a licensed MS- or PhD-level mental health professional experienced in working with persons with dementia and their caregivers. The therapist meets with the AFH owner/operator and staff for four weekly sessions at the AFH. The SEP content includes information about the causes of sleep problems in dementia, and provides staff with assistance in developing customized resident behavioral sleep plans focused on environmental (light and noise), dietary (eliminating caffeine and excessive nighttime fluids), and sleep scheduling (reducing afternoon/ evening napping; consistent, appropriate bed and rising times) factors that are commonly associated with resident nighttime awakenings. A written manual is used.

SUMMARY:
Sleep disturbances are widespread among demented residents of board and care homes and are a leading cause for transfer into nursing homes. This study is a randomized controlled clinical trial to evaluate the efficacy of a 4-week Sleep Education Program (SEP) for demented residents of board and care homes who are experiencing sleep disturbances. Residents of adult family homes (board and care homes with 2-6 residents) will be randomized into SEP or usual care control. Analysis of outcomes will determine whether the SEP is feasible and effective in adult family home settings, and whether the SEP delays transition into higher levels of institutional care.

DETAILED DESCRIPTION:
This study addresses the clinical problem of sleep and nighttime behavioral disturbances in older adults with dementia living in board and care homes. Board and care facilities provide room and board, 24-hour supervision, and assistance with personal care tasks for two or more residents not related to the owner or operator. Many elderly persons who need residential care choose board and care facilities over the alternatives because of their small size and homelike environment.

Adult family homes (AFHs) are small board and care homes with 2-6 residents. Sleep and nighttime behavioral disturbances such as wandering, getting out of bed repeatedly, and day/night confusion are widespread among demented residents of AFHs, and are a leading cause for transfer into nursing homes. However, little is known about how best to treat these problems. Adult family homes vary widely in their type of ownership, staffing schedules, physical environment, resident eligibility criteria, physician access, level of family involvement, and ratio of private/public pay clients. There have been no sleep intervention studies conducted in AFHs, and strategies that have been shown to improve sleep in community-dwelling or nursing home patients may not be feasible or effective in AFH settings. Residents of AFHs have higher rates of functional and health problems that can contribute to sleep disturbances than do community-dwelling patients, and paid caregivers have demanding on-the-job responsibilities and schedules not typically faced by family caregivers. In contrast to skilled nursing facilities, AFH employees often live 24-hours on-site, have limited training in dementia care, and have no licensed health care professionals supervising day-to-day activities. Identification of strategies that could be used as part of a staff educational program to manage sleep and nighttime behavioral disturbances in this unique environment is sorely needed. If successful, such strategies would help residents remain in a less restrictive environment for a longer time, and enhance resident quality of life.

The goal of the project is test the efficacy of a 4-session behavioral intervention for improving sleep and reducing nighttime behavioral disturbances in dementia residents of adult family homes compared to AFH residents in a usual care control condition. This project builds upon previous research conducted by the Principal Investigator showing that brief behavioral interventions can improve sleep of persons with Alzheimer's disease who are living in the community with family caregivers. It applies rigorous methodology to determine whether these interventions are equally feasible and effective in adult family home settings, and whether they delay transition into higher levels of institutional care.

ELIGIBILITY:
Inclusion Criteria:

* Probable or possible AD diagnosis
* Two or more sleep problems on the Sleep Disorders inventory
* Sleep problems occurring three or more times per week
* Living in an Adult Family Home with owner/operator and staff willing to participate

Exclusion Criteria:

* Previously diagnosed primary sleep disorder, e.g. sleep apnea or restless legs syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Actigraphy sleep estimates | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan M McCurry, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States